CLINICAL TRIAL: NCT03970967
Title: A Safety and Effectiveness Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Newly Diagnosed Breast Carcinoma Patients With Distant Metastases
Brief Title: Alpha Radiation Emitters Device for the Treatment of Newly Diagnosed Breast Carcinoma Patients With Distant Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-BRST-01
Record Dates: First submitted 2019-05-23; First posted 2019-06-03 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2022-02

CONDITIONS: Breast Carcinoma; Metastatic Breast Cancer; Invasive Breast Cancer; Distant Metastases.Pathology
Keywords: Breast carcinoma; Metastatic breast cancer; Invasive breast cancer; Alpha radiation; Luminal A; Luminal B; Triple negative; HER2; Breast cancer; Breast metastases
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of radioactive sources [Ra-224 containing stainless-steel 316LVM tubes- (Alpha DaRT seeds)]. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for newly Diagnosed Breast Carcinoma patients with distant metastases

DETAILED DESCRIPTION:
This will be a prospective, open label, single arm, controlled study, assessing the safety and efficacy of diffusing alpha emitters radiation therapy (DaRT) delivered through radioactive sources [Ra-224 containing stainless-steel 316LVM tubes- (Alpha DaRT seeds)] inserted into malignant breast lesions.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Histopathological confirmed invasive breast tumors with no involvement of skin will be treated using DaRT seeds.

The primary effectiveness endpoint of the study is the tumor response to DaRT treatment assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1) 9-11 weeks after DaRT seed insertion.

Safety will be assessed by the cumulative frequency, severity and causality of acute adverse events related to the DaRT treatment of adverse events (AEs) observed including the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathological confirmation of primary (or recurrent) invasive breast carcinoma and distant metastatic disease at diagnosis.
* Target tumor size ≤ 3.0 cm (T1-2b category);
* Morphological type: invasive breast cancer
* Luminal-type A (ER+, PR+, Her2/neu +1), HER+, luminal-type B (ER +/-, PR +/-, Her2/neu+1), or Triple negative breast carcinoma
* Measurable disease according to RECIST v1.1.
* Subjects over 45 years old.
* Subjects' ECOG Performance Status Scale is < 2.
* Subjects' life expectancy more than 6 months.
* Platelet count ≥100,000/mm3.
* International normalized ratio of prothrombin time ≤1.8.
* Creatinine ≤1.9 mg/dL.
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test.
* Subjects are willing to sign an informed consent form.

Exclusion Criteria:

* T4 category with skin involvement.
* Regional lymph node metastases.
* Ductal carcinoma in situ.
* Inflammatory breast carcinoma.
* Patients with pre-irradiation of the breast.
* Acute infection disease.
* The presence of HIV, RW, HbsAg, HCV in the acute stage.
* Pregnancy or lactation.
* Serious competing (somatic) diseases incompatible according to the researcher with brachytherapy.
* Mental illness.
* Patients undergoing immunosuppressive and/or systemic corticosteroid treatment
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator).
* Patients with significant comorbidities that the treating physician deems may conflict with the endpoints of the study (e.g., poorly controlled autoimmune diseases, vasculitis, etc.)
* Subjects not willing to sign an informed consent.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Tumor response to DaRT | 9-11 weeks post DaRT insertion.
  Assessment of the rate of malignant breast tumors response using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1).
Adverse Events | Day 0 - 6 months (+/-14 days)
  Assessment of the frequency, severity and causality of acute adverse events related to the DaRT treatment using the Common Terminology and Criteria for adverse events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Change in tumor volume. | 9-11 weeks after DaRT insertion.
  Assessment of the reduction in tumor volume SUVmax based on CT/PET - CT measured tumor volume.
DaRT seeds placement | Day of insertion.
  Assessment of the DaRT seed placement by localization of the DaRT seed in the tumor using CT imaging.
Change in quality of life: EORTC-QLQ-C30 | Day 0, 30, 70, 6 months (+/-14 days).
  Assessment of patient reported health-related Quality of Life (QoL) outcomes after DaRT treatment, using QoL questionnaires EORTC-QLQ-C30. Scale range in score from 0 (best) to 100(worst).
Progression free survival | 6 months (+/-14 days).
  Time elapsed from response to disease progression.
Pathological remissions. | 12 weeks after DaRT seed insertion.
  Assessment of (complete) pathological remissions using histopathology examination
Abscopal effects. | 9-11 weeks after DaRT insertion.
  Assessment of abscopal effects on existing distant metastases based on PET-CT measured tumor volume.
Change in quality of life: BR23 | Day 0, 30, 70, 6 months (+/-14 days).
  Assessment of patient reported health-related Quality of Life (QoL) outcomes after DaRT treatment, using QoL questionnaires BR23. Scale range in score from 0 (best) to 100(worst).
Abscopal effects | 9-11 weeks after DaRT insertion.
  Assessment of abscopal effects on existing distant metastases based on PET-CT measured SUVmax decrease compared to the primary measurement (the baseline measurement).

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr Obukhov, Principal Investigator — A. Tsyb Medical Radiological Research Centre, (A. Tsyb MRRC), Obninsk, Russia
Locations (1):
- A. Tsyb Medical Radiological Research Center, Obninsk, Kaluga Oblast, Russia

IPD SHARING:
Plan to Share IPD: No